CLINICAL TRIAL: NCT04262115
Title: Feasibility and Acceptability of Morning Versus Evening Exercise for Adults With Overweight and Obesity: A Randomized Pilot Study
Brief Title: Morning Versus Evening Exercise for Adults With Overweight and Obesity
Acronym: TIC-TOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-2676
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Overweight and Obesity
Keywords: exercise; physical activity; weight loss
MeSH Terms: conditions — Overweight; Obesity; Motor Activity; Weight Loss

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AM-EX (Experimental): Participants in this group will be prescribed morning aerobic exercise.
  Interventions: Behavioral: AM-EX
- PM-EX (Experimental): Participants in this group will be prescribed evening aerobic exercise.
  Interventions: Behavioral: PM-EX

INTERVENTIONS:
Behavioral: AM-EX — AM will be instructed to perform 2000 kcal/wk of moderate to vigorous intensity aerobic exercise between the hours of 6 and 10 AM.
  Arms: AM-EX
Behavioral: PM-EX — PM will be instructed to perform 2000 kcal/wk of moderate to vigorous intensity aerobic exercise between the hours of 3 and 7 PM.
  Arms: PM-EX

SUMMARY:
The purpose of this pilot study is to determine the feasibility and acceptability of randomizing adults with overweight and obesity to an exercise intervention of either prescribed morning aerobic exercise (AM-EX) or prescribed evening aerobic exercise (PM-EX) progressing to 2000 kcal/wk.

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine the feasibility and acceptability of randomizing adults with overweight and obesity to an exercise intervention of either prescribed morning aerobic exercise (AM-EX) or prescribed evening aerobic exercise (PM-EX) progressing to 2000 kcal/wk. Specifically, the purpose of this study is to assess recruitment, retention, and adherence to the exercise interventions.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male
* Age 18-55 years
* Body Mass Index 25-40 kg/m2
* Physically inactive: defined as self-reporting <150 minutes per week of physical activity at moderate intensity or greater on a regular basis over the past 3 months.
* No self-report of acute or chronic disease (cardiovascular disease (CVD), diabetes, gastrointestinal disorders and orthopedic problems in particular)
* No plans to relocate within the next 6 months
* No plans for extended travel (> 1weeks) within the next 6 months
* No nicotine use
* Live or work within 30 minutes of the AHWC (exceptions may be made at the discretion of the Study PI on a case by case basis for highly motivated subjects).
* Capable and willing to give informed consent, understand exclusion criteria, accept the randomized group assignment, and complete outcome measures.
* Own a smartphone and willing to download and use text messaging for meal intake and other related assessments.
* Have a primary care physician (or are willing to establish care with a primary care physician prior to study enrollment) to address medical issues which may arise during screening or study procedures/interventions.
* For Females

  * Not currently pregnant or lactating
  * Not pregnant within the past 6 months
  * Not planning to become pregnant in the next 6 months; sexually active women of childbearing potential may be enrolled if they have had a tubal ligation or use a reliable means of contraception

Exclusion Criteria:

* Diastolic blood pressure > 100 mm HG or systolic blood pressure > 160 mm HG.
* Resting heart rate >100
* Diabetes (fasting glucose ≥126 mg/dL or Hemoglobin A1C ≥6.5%)
* Undiagnosed hypo- or hyper-thyroidism (TSH outside of the normal range) or history of uncontrolled thyroid disorder. History of thyroid disease or current thyroid disease treated with a stable medication regimen for at least 6 months is acceptable.
* Hematocrit, white blood cell count or platelets significantly outside the normal reference range.
* Triglycerides > 400 mg/dL
* LDL cholesterol >200 mg/dL
* Abnormal resting electrocardiogram (ECG): serious arrhythmias, including multifocal PVC's, frequent PVC's (defined as 10 or more per min), ventricular tachycardia (defined as runs of 3 or more successive PVC's), or sustained atrial tachyarrhythmia; 2nd or 3rd degree A-V block, QTc interval > 480 msec or other significant conduction defects.
* Presence or history of any metabolic or chronic health problems which would affect appetite, food intake, energy metabolism, or ability to optimally participate in the exercise component including: CVD, peripheral vascular disease, cerebrovascular disease, significant cardiac arrhythmias or cardiac valve disease, diabetes, uncontrolled hyper- or hypothyroidism, uncontrolled hypertension, cancer (within the last 5 years, except skin cancer or other cancers considered cured with excellent prognosis), HIV infection, significant gastrointestinal disorders (described below), significant pulmonary disorders (described below), significant renal, musculoskeletal, neurologic, hematologic, or psychiatric disease.
* Significant gastrointestinal disorders including: chronic malabsorptive conditions, peptic ulcer disease, Crohn's disease, Ulcerative Colitis, chronic diarrhea, or active gallbladder disease.
* Significant pulmonary disorders including: chronic obstructive pulmonary disease (COPD), interstitial lung disease, cystic fibrosis, or uncontrolled asthma.
* Symptoms suggestive of CVD: chest pain, shortness of breath at rest or with mild exertion, syncope.
* Regular use of prescription or over-the-counter medications known to significantly impact appetite, weight, sleep, or energy metabolism (e.g. appetite suppressants, lithium, stimulants, anti-psychotics, tricyclic antidepressants)
* Regular use of systemic steroids (other than Oral Contraceptive Pills).
* Regular use of obesity pharmacotherapeutic agents within the last 6 months.
* Previous obesity treatment with surgery or weight loss device, except: (1) liposuction and/or abdominoplasty if performed > 1 year before screening, (2) lap banding if the band has been removed > 1 year before screening, (3) intragastric balloon if the balloon has been removed > 1 year before screening (4) duodenal-jejunal bypass sleeve, if the sleeve has been removed > 1 year before screening or 5) AspireAssist or other endoscopically placed weight loss device if the device has been removed > 1 year before screening.
* Current alcohol or substance abuse
* Irregular sleep/wake patterns that may hinder ability to consistently exercise at a certain time of day (e.g. night shift-work, swing shifts, etc)
* Currently dieting or planning to alter diet during the exercise intervention
* Nicotine use (past 6 months)
* History of clinically diagnosed eating disorders including anorexia nervosa, bulimia, binge eating disorder. Pattern of response on the QEWP-5 suggestive of possible binge eating disorder or bulimia will require further assessment by the Study MD to determine if it is appropriate for the subject to participate in the study.
* Current severe depression or history of severe depression within the previous year, based on DSM-IV-TR criteria for Major Depressive Episode. Score > 18 on BDI will require further assessment by the Study MD to determine if it is appropriate for the subject to participate in the study.
* History of other significant psychiatric illness (e.g. psychosis, schizophrenia, mania, bipolar disorder) which in the opinion of the Study MD would interfere with ability to adhere to dietary or exercise interventions.
* Currently participating in or planning to participate in any formal weight loss or physical activity programs or clinical trials.
* Weight loss >5% in past 3 months for any reason except post-partum weight loss, weight gain >% in past 3 months requires assessment by PI to determine reason for weight gain and if it is appropriate for the subject to participate in the study.
* Weight loss of >50 lbs in past 3 years for any reason except post-partum weight loss.

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of Recruitment (Number of contacts) | End of enrollment (estimated between 6 and 12 months)
  Feasibility of recruitment will be evaluated by the number of people who contact study staff expressing interest in the study
Feasibility of Recruitment (eligibility rate) | End of enrollment (estimated between 6 and 12 months)
  Feasibility of recruitment will be evaluated by calculating the number of volunteers who contact study staff to express interest in participation, the eligibility rate (number eligible divided by total volunteers)
Feasibility of Recruitment (enrollment rate) | End of enrollment (estimated between 6 and 12 months)
  Feasibility of recruitment will be evaluated by calculating the enrollment rate (number enrolled divided by the number of total volunteers)
Adherence to Exercise Intervention (session attendance) | Baseline to 15 weeks (reported at Week 15)
  Adherence will be calculated as (number of sessions attended/number of sessions prescribed)
Adherence to Exercise Intervention (kcal adherence) | Baseline to 15 weeks (reported at Week 15)
  Adherence will be calculated as (number of kcals prescribed/ number of kcals of exercise completed)

SECONDARY OUTCOMES:
Weight Change (kg) | Baseline to 15 weeks
  Body weight will be measured at baseline and weeks 4, 8, 12, and 15 using a digital scale accurate to ±0.1 kg
Physical Activity Change (min/d) | Baseline to 15 weeks
  Physical activity will be measured using the ActivPAL v4
Meal Timing Change (clock time of first meal) | Baseline to 15 weeks
  Meal timing will be assessed using digital photography paired with a date and time stamp (time of first meal)
Meal Timing Change (clock time of last meal) | Baseline to 15 weeks
  Meal timing will be assessed using digital photography paired with a date and time stamp (time of last meal)
Sleep Timing Change (mid-point of sleep) | Baseline to 15 weeks
  Mid-point of sleep will be measured using the Actiwatch 2 (starting sleep time + (sleep duration/2))

CONTACTS AND LOCATIONS:
Overall Officials: Seth A Creasy, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No